CLINICAL TRIAL: NCT05203159
Title: The Effect of Ocean Sound on Physiological Parameters, Pain and Comfort Level In Premature Retinopathy Examination: A Randomized Controlled Study
Brief Title: The Effect of Ocean Sound In Premature Retinopathy Examination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Gülay ARSLAN, Lecturer, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 12345
Record Dates: First submitted 2021-12-13; First posted 2022-01-24 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Premature Retinopathy; Pain
MeSH Terms: conditions — Retinopathy of Prematurity; Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ocean sound (Experimental): The group that will listen to the ocean sound
  Interventions: Other: Ocean sound
- control group (Active Comparator): The group that will not listen to sound
  Interventions: Other: Routine

INTERVENTIONS:
Other: Ocean sound — The experimental group will listen to ocean sound, starting at the 1st minute before the ROP examination and ending at the 5th minute after the ROP examination.
  Arms: ocean sound
Other: Routine — No sound will be played before, during and after the ROP examination.
  Arms: control group

SUMMARY:
Purpose: It was planned as a randomized controlled experiment in order to evaluate the effectiveness of the ocean sound on pain, comfort and physiological parameters in the NICU, Retinopathy of Prematurity (ROP) examination.

Design: This is single-center. randomized controlled trial, double blind, parallel.

Hypotheses:

H0a: There is no difference between the pain levels (scale score) of premature babies in the control group and the ocean sound group.

H0b: There is no difference between the comfort levels (scale score) of premature babies in the control group and the ocean sound group.

H0c: There is no difference between the physiological parameters of the premature babies in the control group and the ocean sound group.

H1a: There is a difference between the pain levels (scale score) of premature babies in the control group and the ocean sound group.

H1b: There is a difference between the comfort levels (scale score) of premature babies in the control group and the ocean sound group.

H1c: There is a difference between the physiological parameters of the premature babies in the control group and the ocean sound group.

Method:

The population of the research will be preterm babies who are treated at Necmettin Erbakan University Meram Medical Faculty NICU and will have their first ROP examination.

Premature babies to be included in the study will be assigned to two study groups using the quadruple balanced block randomization method created in the computer environment according to their gestational age.

In the study, the baby information form, Premature Baby Pain Profile Scale-Revised Form (PIPP-R), and Premature Baby Comfort Scale (PBIC) created by the researcher by scanning the literature will be used.

Data will be collected by researcher GA. Infants who meet the criteria for inclusion in the study will be selected from the infants who are planned to undergo an ROP examination, and written and verbal consent will be obtained from the families by explaining the purpose of the study before the application.

The information contained in the "Baby Information Form" will be obtained from the nurse observation form and patient files. On the day of the ROP examination, babies who meet the inclusion criteria before the procedure will be recorded outside the incubator with a video recorder in the room where the ROP examination will be performed (a room with 45-50 dB sound). Two minutes before the ROP, the baby will be monitored and physiological parameters will be recorded, and one minute before the ROP, the experimental group will start to listen to the ocean sound (Video recordings will be evaluated by two experts, PIPP-R and PBIC). After the necessary disinfection process is done, the voice recorder will be placed in the incubator at a distance of 20 cm from the baby's head and the sound level will be adjusted to an average of 55 decibels. The examination will begin with the placement of the speculum in the eye. The duration of the examination varies according to the visibility of the retinal vascularity, and the examination will end with the removal of the speculum from the eye. Ocean Sound Group; The ocean sound recording will continue to be played during the ROP examination. Control Group; No sound will be played before, during and after the ROP examination.

Physiological parameters will be recorded at the 1st and 5th minutes after the procedure. (Video recordings will be evaluated by two experts for PIPP-R and PBIC). Video recording will be stopped.Ocean Sound Group;The ocean sound recording will be played at the 5th minute after the ROP inspection. Control Group; No sound will be played before, during and after the ROP examination.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age ≤32 weeks
* Birth Weight ≤2000 grams
* Receiving babies that the clinician following the baby deems at risk for the development of ROP
* Receiving babies who will have their first ROP examination
* No sedative, opioid and anticonvulsant medication given before/during the examination
* Parents do not have diagnosed mental or mental problems and agree to participate in the research.

Exclusion Criteria:

* Presence of a condition that interferes with pain assessment (intracranial hemorrhage, neuro-motor developmental delay, etc.)
* Diagnosed hearing loss
* Performing a different painful procedure before the ROP (one hour)
* Being connected to a mechanical ventilator
* Congenital hearing problems in family members

Ages: 28 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2021-11-25 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-06-13 (Actual)

PRIMARY OUTCOMES:
Heart Rate | The measurement will start 2 minutes before the ROP examination and will end 5 minutes after the ROP examination (the examination ends with the removal of the speculum).
  A pulse oximeter device will be used.
Oxygen Saturation | The measurement will start 2 minutes before the ROP examination and will end 5 minutes after the ROP examination (the examination ends with the removal of the speculum).
  A pulse oximeter device will be used.
Premature Baby Pain Profile Scale-Revised Form (PIPP-R) | The measurement will start 2 minutes before the ROP examination and will end 5 minutes after the ROP examination (the examination ends with the removal of the speculum).
  The PIPP-R is a Likert-type scale. In scoring the scale, items related to physiological and behavioral elements are scored as 0, 1, 2, 3, reflecting the difference between the values at baseline and during the procedure in each variable. Contextual items (behavioral status and CI) are scored as 3, 2, 1, 0 only at the beginning of the pain assessment (before touching the baby). According to the PIPP-R, the baby's pain is evaluated over the total score. Accordingly, the highest score that can be obtained from the PIPP-R scale for preterm newborns is 21 and 18 for term newborns.
Premature Infant Comfort Scale (PBIC) | The measurement will start 2 minutes before the ROP examination and will end 5 minutes after the ROP examination (the examination ends with the removal of the speculum).
  The scale was prepared in a 5-point Likert type consisting of 7 sub-dimensions and 35 items. The scale is a multidimensional scale used to evaluate behavioral and psychological comfort and pain. It evaluates 7 parameters such as Alertness, Calmness/Agitation, Breathing Status or Crying, Physical Movement, Muscle Tone, Facial Movements and Average Heart Rate.As the scores obtained from the scale increase, the baby's comfort level decreases. While 35 points indicates the lowest comfort level, 7 points indicates the highest comfort level.

CONTACTS AND LOCATIONS:
Locations (1):
- Necmettin Erbakan University Meram Medical Faculty Hospital Neonatal Intensive Care Unit, Konya, Meram/Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No